CLINICAL TRIAL: NCT02804308
Title: Effectiveness of Physical Training on Body Composition, Physical Activity Level and Quality of Life of Postmenopausal Women Undergoing Treatment for Breast Cancer With Aromatase Inhibitors: The Randomized Clinical Trial.
Brief Title: Combined Training on Body Composition of Postmenopausal Women Undergoing Treatment for Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Thais Reis Silva de Paulo, masters degree, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: CAAE46727715100005402
Record Dates: First submitted 2016-06-10; First posted 2016-06-17 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2015-03

CONDITIONS: Breast Cancer; Aromatase Inhibitors; Postmenopausal
Keywords: Combined Training; Breast Cancer; Body Composition; Postmenopausal Women; Aromatase Inhibitors; Quality of life
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group Control with breast cancer and without breast cancer (No Intervention): Stretching exercises, lasting 40 minutes each session, 2 times a week for nine months
- Combined Training with breast cancer and without breast cancer (Experimental): Combined Training: 36 weeks duration, 3 times a week on nonconsecutive days. The combined training program lasts 70 minutes per session, with 40 minutes of resistance training and 30 minutes of aerobic training.
  Interventions: Behavioral: Combined Training

INTERVENTIONS:
Behavioral: Combined Training
  Arms: Combined Training with breast cancer and without breast cancer

SUMMARY:
Breast cancer is a multifactorial disease affecting women, and one of the treatments for its healing and survival is hormone therapy. Aromatase inhibitors are third-generation drugs that promote lower chance of metastasis, but their side effects include the loss of bone mineral density and increased fat percentage. In this way, the Combined Training (combined resistance and endurance training) may be an interesting strategy to minimize the side effects of aromatase inhibitors, providing better quality of life, survival and changes in body composition.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal, defined by the absence of periods for the past 12 months;
* Breast cancer diagnosis stages 1 to 3;
* The adjuvant treatment for breast cancer and / or neoadjuvant aromatase inhibitors
* No abnormalities on screening physical or any health problems that contraindicate study participation;
* No contraindications for treadmill testing or entry into a training program, including any of the following:
* Myocardial infarction within the past 6 months
* Pulmonary edema
* Myocarditis Pericarditis
* Unstable angina
* Pulmonary embolism or deep vein thrombosis
* Uncontrolled hypertension (i.e., blood pressure > 200/100 mm Hg)
* Uncontrolled arrhythmia
* No significant mental illness
* Have medical certificate to perform exercise testing and participate in combined training
* Able to answer Questionnaires
* No concurrent participation in any other organized exercise program;
* Live in Presidente Prudente
* Sign the consent form and formal clarification for participation in the study.

Exclusion Criteria:

* Accumulating 3 unexcused absences or 4 consecutive unexcused absences during the month.

Ages: 50 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2015-08; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Chance from Body composition at 9 months assessment by bone densitometry (Dual-energy x-ray absorptiometry), using the equipment model GE Lunar - DPX-NT | At baseline, 3, 6 and 9 months timepoint

SECONDARY OUTCOMES:
Quality of life assessed via the questionnaire EORTC (European Organization for Research and Treatment of Cancer Quality of Life Questionnarie). | At baseline, 3, 6 and 9 months timepoint
Bone mineral density (total, spine and femur) in these participants by bone densitometry (Dual-energy x-ray absorptiometry), using the equipment model GE Lunar - DPX-NT. | At baseline, 3, 6 and 9 months timepoint
Serum levels of glucose in these participants measured by enzymatic colorimetric kit processed in Autohumalyzer A5 | At baseline, 3, 6 and 9 months timepoint
Serum levels of C-reactive protein (CRP) in these participants measured by enzymatic colorimetric kit processed in Autohumalyzer A5 | At baseline, 3, 6 and 9 months timepoint
Serum levels of total cholesterol and fractions in these participants measured by enzymatic colorimetric kit processed in Autohumalyzer A5. | At baseline, 3, 6 and 9 months timepoint
Serum levels of triacylglycerol in these participants measured by enzymatic colorimetric kit processed in Autohumalyzer A5 | At baseline, 3, 6 and 9 months timepoint
Serum of osteocalcin and the carboxyterminal telopeptides of collagen type I (CTX) measured at Serum CrossLaps Assay | At baseline, 3, 6 and 9 months timepoint
Physical Activity of accelerometer motion sensor type triaxial Actigraph brand, mode GT3X. | At baseline, 3, 6 and 9 months timepoint
The perception of pain is measured by Pain Brief Questionnaire (PBQ | At baseline, 3, 6 and 9 months timepoint
VO2max by test of submaximal effort | At baseline, 3, 6 and 9 months timepoint
Responsiveness on body composition by bone densitometry (Dual-energy x-ray absorptiometry). | At baseline, 3 and 6 months timepoint
Responsiveness on habitual physical activity by accelerometer motion sensor type triaxial Actigraph brand, mode GT3X (Actigraph LLC, Pensacola, FL). | At baseline, 3 and 6 months timepoint
Use time of aromatase inhibitor and the response to combined training in the variables of body composition and level of physical activity by bone densitometry (GE Lunar - DPX-NT) and accelerometer motion sensor type triaxial Actigraph brand, mode GT3X | At baseline, 3 and 6 months timepoint
Self reported Drug consumption questionnaire | At baseline, 3, 6 and 9 months timepoint

CONTACTS AND LOCATIONS:
Overall Officials: Ismael F Freitas Junior, Doctor, Study Director — UPECLIN HC FM Botucatu Unesp

REFERENCES:
- [Derived] Felipe J, Viezel J, Reis AD, da Costa Barros EA, de Paulo TRS, Neves LM, Junior IFF. Relationship of different intensities of physical activity and quality of life in postmenopausal women. Health Qual Life Outcomes. 2020 May 6;18(1):123. doi: 10.1186/s12955-020-01377-1. PMID 32375779